CLINICAL TRIAL: NCT03344796
Title: A Real-time, Cost-effective, Accurate UV Measurement and Sun Protection System to Prevent and Reduce the Incidence of Sunburn in High-risk Consumers
Brief Title: UV Exposure Assessed With Wearable Sensor and Sun Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, June Robinson, Primary Investigator, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STU00205910; R44CA224658 (NIH)
Record Dates: First submitted 2017-10-26; First posted 2017-11-17 (Actual); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Sunburn, Erythema; Sun Protection
Keywords: Skin Cancer; Sunburn, erythema; UV Exposure, Sunburn; Wearable UV Device
MeSH Terms: conditions — Sunburn; Erythema; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: Cohort study 1 is parallel and randomized Cohort Study 2 is a single group study with comparison of the participants' reported sunburns prior to intervention and during the intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: cohort study 1 and 2 were masked. Each participant was identified by a study number assigned in REDCap
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Focus Group (No Intervention): 32 subjects
  Focus group: It is expected that each participant will provide comments during the 2 hours of the focus group. It will take about one month to enroll the subjects. The audio files should be transcribed and the analysis completed in 60 days. The analysis will determine enablers and barriers to sun protected outdoor activities and determine strategies for achieving sun protected outdoor activities. Baseline knowledge of sun protection performed prior to and at end of focus group.
- Usability testing (No Intervention): 10 subjects
  Usability test with structured interview: Each participant will use the sensor for 14 days and transmit data with the app installed on their mobile phone. It will take about one month to enroll the subjects. The analysis of the structured interview is completed in one week. Baseline knowledge of sun protection performed prior to and at end of usability test.
- Cohort Study 1-Arm 1 (Active Comparator): 31 subjects
  First cohort study: It is expected that melanoma survivors will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will be randomized in Arm 1 to receive a survey item inviting selection of strategies to achieve sun-protected outdoor activities (structured goal attainment). Baseline knowledge of sun protection performed prior to and at end of intervention.
  Interventions: Behavioral: Goal attainment
- Structured Interviews (No Intervention): 20 young adults, ages 18-39 will participate in structured interviews to determine their barriers and enablers of sun exposure and sun protection. Eligible subjects will have at least one hour a day outdoors with 30 minutes of the hour being consecutive. It will take about 3 months to enroll the subjects. The audio files will be transcribed and analysis completed in 60 days. Baseline knowledge of sun protection will be performed prior to and after structured interviews.
- Cohort Study 2 (No Intervention): Second cohort study: 42 young adult participants will recall the number of sunburns experienced in the 28 days prior to enrolling in the study. Then, the same young adult participants will wear the UV sensor daily for 28 summer days. Participants will receive a warning on their mobile phone if the UV dose approaches the dose anticipated to cause sunburn in unprotected skin. Participants will record the number of days in which they get a sunburn. Baseline knowledge of sun protection performed prior to and at end of study.
- Cohort Study 1- Arm 2 (Active Comparator): 29 subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will be randomized in Arm 2 to submit a free text description of their strategy (unstructured goal attainment). Baseline knowledge of sun protection performed prior to and at end of intervention.
  Interventions: Behavioral: Goal attainment

INTERVENTIONS:
Behavioral: Goal attainment — After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
  Arms: Cohort Study 1- Arm 2; Cohort Study 1-Arm 1

SUMMARY:
The goal is to prevent ultraviolet light (UV) overexposure by providing consumers with relevant, easy-to-access, specifically actionable information. This research proposal will develop a UV protection system consisting of an automated real-time counseling framework and a personal dosimeter that overcomes barriers to consumer adoption. These new, wearable sensors take the form of small (< 1 cm), thin (<0.1 mm), lightweight (<0.1 g), battery-free "stickers" that are fundamentally differentiated from other wearable electronics in their modes of use, cost structures and accuracy.

DETAILED DESCRIPTION:
The proposed work is to refine and validate a UV protection system based on a dosimeter "sticker." The key innovations of the system are automated personalized intervention messaging triggered by the exposure levels measured by a novel charge accumulation device applied to ultraminiaturized circuit forms. The research will validate the system's accuracy and acceptability to users, refine the device, and prove its robustness and efficacy in real world use cases. Focus groups and structured interviews will develop sun protection strategies to be communicated by text messages to participants. Successful completion of the research will yield a system to prevent excessive UV exposure and sunburn, thus reducing the incidence of skin cancer by equipping large numbers of general-population consumers and at-risk people to practice digitally-informed healthy sun behavior.

ELIGIBILITY:
Cohort Study 1:

Inclusion Criteria:

1. history of Stage 0 to IIB melanoma treated within the last five years, age 18-70 years old
2. have a smartphone
3. familiarity with use of mobile apps
4. have skin type 1-3
5. willing to wear the sensor and able to transmit data which requires Wi-Fi in the home
6. Come to the Chicago campus of the medical school

Exclusion Criteria:

-

Cohort Study 2: Young adults with sun sensitive skin

Inclusion Criteria:

1. history of sun sensitive skin, skin type 1-3
2. have a smartphone and willing to use the UV guard application on the smartphone
3. reliable wireless internet connection to complete daily surveys
4. willing to wear the sensor for 28 days and transmit data and complete daily surveys
5. willing to receive SMS text messages on their personal phone and potentially sync sensor to personal phone using Bluetooth
6. If weather permits, person will spend at least one hour outdoors each day, with at least 30 minutes of that hour being consecutive between the hours of 8 AM and 5 PM

Exclusion Criteria:

1. unable to speak English
2. lacking a secure Internet connection or very little experience with smartphones and mobile applications .
3. unable to walk inside and outside independently
4. unable to be outdoors for at least one hour each day (weather permitting)
5. unable to be outdoors for 30 consecutive minutes a day between 8 AM and 5 PM.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-06-30 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: June K. Robinson, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine Department of Dermatology, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Robinson JK, Durst DA, Gray E, Kwasny M, Heo SY, Banks A, Rogers JA. Sun exposure reduction by melanoma survivors with wearable sensor providing real-time UV exposure and daily text messages with structured goal setting. Arch Dermatol Res. 2021 Oct;313(8):685-694. doi: 10.1007/s00403-020-02163-1. Epub 2020 Nov 13. PMID 33185716
- [Result] Stump TK, Aspinwall LG, Gray EL, Xu S, Maganti N, Leachman SA, Alshurafa N, Robinson JK. Daily Minutes of Unprotected Sun Exposure (MUSE) Inventory: Measure description and comparisons to UVR sensor and sun protection survey data. Prev Med Rep. 2018 Jul 24;11:305-311. doi: 10.1016/j.pmedr.2018.07.010. eCollection 2018 Sep. PMID 30116702
- [Derived] Robinson JK, Patel S, Heo SY, Gray E, Lim J, Kwon K, Christiansen Z, Model J, Trueb J, Banks A, Kwasny M, Rogers JA. Real-Time UV Measurement With a Sun Protection System for Warning Young Adults About Sunburn: Prospective Cohort Study. JMIR Mhealth Uhealth. 2021 May 6;9(5):e25895. doi: 10.2196/25895. PMID 33955844

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for the overall study: June 30, 2018 - June 30, 2020. Participants for the first cohort (cohort 1) were recruited using the Enterprise Data Warehouse of Northwestern University, which searches the electronic medical records of Northwestern Medicine for eligible participants.
  Participants for the second cohort (cohort 2) were recruited by posting electronic announcements on college websites and high school alumnae organizations in the Midwestern and Southeastern United States.
Pre-assignment Details: After subject meets eligibility requirements and is enrolled they are assigned to an arm without a run-in or wash-out.
Groups:
- Focus Group: 32 subjects
  Focus group: It is expected that each participant will provide comments during the 2 hours of the focus group. It will take about one month to enroll the subjects. The audio files should be transcribed and the analysis completed in 60 days. The analysis will determine enablers and barriers to sun protected outdoor activities and determine strategies for achieving sun protected outdoor activities.
- Usability Testing: 10 subjects
  Usability test with structured interview: Each participant will use the sensor for 14 days and transmit data with the app installed on their mobile phone. It will take about one month to enroll the subjects. The analysis of the structured interview is completed in one week.
- Cohort Study 1- Arm 1: 31 subjects
  First cohort study: It is expected that each of 31 melanoma survivors will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will receive a survey item inviting selection of strategies to achieve sun-protected outdoor activities (structured goal attainment) Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will receive structured (select strategies from a list of 7 items)
- Cohort Study 1 Arm 2: Each of 29 melanoma survivors in arm 2 will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects in both arms will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants in arm 2 will be randomized to submit a free text description of their strategy (unstructured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to unstructured (submit a free text description of a strategy) goal attainment.
- Structured Interviews: 20 young adults, ages 18-39 will participate in structured interviews to determine their barriers and enablers of sun exposure and sun protection. Eligible subjects will have at least one hour a day outdoors with 30 minutes of the hour being consecutive. It will take about 3 months to enroll the subjects. The audio files will be transcribed and analysis completed in 60 days.
- Cohort Study 2: Second cohort study: 42 young adults will wear the sensor and transmit data for 28 days in summer 2020.
Period: Overall Study
Arm/Group | Focus Group | Usability Testing | Cohort Study 1- Arm 1 | Cohort Study 1 Arm 2 | Structured Interviews | Cohort Study 2
Started | 32 | 10 | 31 | 29 | 20 | 42
Completed | 32 | 10 | 31 | 29 | 20 | 40 (Daily online survey data was not completed by 2 participants.)
Not Completed | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Cohort Study 1 Arm 1: 31 subjects
  First cohort study: It is expected that each of 60 melanoma survivors in arms 1 + 2 will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects in both arms will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants in arm 1 will be randomized to receive a survey item inviting selection of strategies to achieve sun-protected outdoor activities (structured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
- Cohort Study 1 Arm 2: 29 subjects
  First cohort study: It is expected that each of 29 melanoma survivors in arm 2 will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects in both arms will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants in arm 2 will be randomized to submit a free text description of their strategy (unstructured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
- Cohort Study 2: Second cohort study: 42 young adults will recall the number of days with a sunburn in the 28 days before the intervention. Then, the same young adults will wear the UV sensor daily for 28 days in summer 2020. The UV sensor will provide an alert when the UV exposure approaches the dose expected to produce a sunburn. Participants will report sunburns daily during the 28 days of the intervention.
- Total: Total of all reporting groups
Arm/Group | Focus Group | Usability Testing | Cohort Study 1 Arm 1 | Cohort Study 1 Arm 2 | Structured Interviews | Cohort Study 2 | Total
Number analyzed (Participants) | 32 | 10 | 31 | 29 | 20 | 42 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 25 | 10 | 25 | 24 | 20 | 42 | 146
  >=65 years | 7 | 0 | 6 | 5 | 0 | 0 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.4 (11.5) | 24.3 (3.2) | 59.3 (12.5) | 58.8 (10.2) | 21.2 (1.4) | 22.6 (4.5) | 48.2 (15.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 5 | 18 | 18 | 10 | 28 | 96
  Male | 15 | 5 | 13 | 11 | 10 | 14 | 68
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 1 | 0 | 0 | 1 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 30 | 9 | 31 | 29 | 18 | 36 | 153
  More than one race | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 32 | 10 | 31 | 29 | 20 | 42 | 164
Knowledge of Sun Protection [Mean (Standard Deviation); unit: units on a scale] — 9 item scale (Minimum= 9, Maximum=18) Total range is9-18. Higher value is better knowledge and a better outcome.
  units on a scale | 12 (1.7) | 13 (3.1) | 17 (2.3) | 18 (1.9) | 11 (1.4) | 11 (2.1) | 14 (2.1)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Wearing UV Sensor and Receiving Text Messages
Description: Online system usability 6 item scale (Likert 7 items range from strongly disagree to strongly agree Minimum value 6, maximum value 42, higher score better outcome
Time Frame: cohort study 1 (arms 1 and 2) at end of 21 days, cohort study 2 (only one arm) at end of 28 days
Population: Focus groups and structured interviews did not have data collected for acceptability of wearing the UV sensor and receiving text messages.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cohort Study 1 Arm1: 31 subjects
  First cohort study: It is expected that each of 60 melanoma survivors in arms 1+2 will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will be randomized to receive a survey item inviting selection of strategies to achieve sun-protected outdoor activities (structured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
- Cohort Study 1 Arm 2: 29 subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will be randomized tosubmit a free text description of their strategy (unstructured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
Arm/Group | Usability Testing | Cohort Study 1 Arm1 | Cohort Study 1 Arm 2 | Cohort Study 2
Number analyzed (Participants) | 10 | 31 | 29 | 42
score on a scale | 22 (3.5) | 39.1 (6.2) | 40.1 (5.3) | 40.6 (2.9)
Statistical Analysis 1: Comparison: Cohort Study 1 Arm1 vs Cohort Study 1 Arm 2 vs Cohort Study 2; Test type: Superiority; p < 0.01, Chi-squared

2. Secondary Outcome: Sun Exposure in Participants With Structured vs Unstructured Goal Setting
Description: Change in daily UV exposure recorded by UV sensor (J/m^2/day) between period prior to and after goal setting among melanoma survivors
Time Frame: 21 days
Population: UV exposure as recorded by the UV sensor in J/m^2 per day from period 1 (prior to goal setting) to period 2 (after goal setting) only applies to cohort study 1. The other study arms focus group, usability test, unstructured interview and Cohort study 2 did not have data collected.
Measure: Least Squares Mean (Standard Error); unit: J/m^2/day
Groups:
- Cohort Study 1 Arm 1: 31 subjects
  First cohort study: It is expected that melanoma survivors in arm 1 will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will be randomized to receive a survey item inviting selection of strategies to achieve sun-protected outdoor activities (structured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
- Cohort Study 1 Arm 2: Subjects in arm 2 will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. 29 participants in arm 2 will be randomized to submit a free text description of their strategy (unstructured goal attainment).
Arm/Group | Cohort Study 1 Arm 1 | Cohort Study 1 Arm 2
Number analyzed (Participants) | 31 | 29
J/m^2/day | 399.9 (10.6) | 196.8 (129.1)
Statistical Analysis 1: Comparison: Cohort Study 1 Arm 1 vs Cohort Study 1 Arm 2; Test type: Superiority; p < 0.001, Chi-squared, Corrected

3. Other Pre Specified Outcome: Participant Reported Sunburns Prior to Intervention and During the Intervention
Description: Young adult participants with sun sensitive skin reported sunburns in the 28 days prior to the intervention and during the 28 days of the intervention.
Time Frame: 56 days
Population: This is a single arm study for cohort 2. Data on sunburns was not collected for the other arms.
Measure: Number; unit: participants
Groups:
- Participant Reported Sunburns: Young adults with sun sensitive skin reported the number of days with a sunburn for the 28 days prior to the intervention. Then participants reported daily sunburn during the study.
Arm/Group | Participant Reported Sunburns
Number analyzed (Participants) | 42
participants
  Sunburns prior to intervention | 30
  Sunburns during intervention | 18
Statistical Analysis 1: Comparison: Participant Reported Sunburns; Test type: Superiority; p < 0.01, Chi-squared

4. Other Pre Specified Outcome: Knowledge of Sun Protection
Description: Knowledge of sun protection using the scale after completing focus group after completing an arm of the study. The same scale was administered at baseline for each arm.
  9 item scale (Minimum= 9, Maximum=18) Total range is 9-18. Higher value is better knowledge and a better outcome.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Cohort Study 1-Arm 1: 31 subjects
  First cohort study: It is expected that each of 31 melanoma survivors will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will be randomized in Arm 1 to receive a survey item inviting selection of strategies to achieve sun-protected outdoor activities (structured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
- Cohort Study 1- Arm 2: Subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will be randomized in Arm 2 to submit a free text description of their strategy (unstructured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
Arm/Group | Focus Group | Usability Testing | Cohort Study 1-Arm 1 | Cohort Study 1- Arm 2 | Structured Interviews | Cohort Study 2
Number analyzed (Participants) | 32 | 10 | 31 | 29 | 20 | 40
score on a scale | 13.2 (0.2) | 13.1 (0.5) | 17.9 (1.1) | 17.1 (1.2) | 12.2 (0.4) | 14.3 (0.6)
Statistical Analysis 1: Comparison: Focus Group vs Usability Testing vs Cohort Study 1-Arm 1 vs Cohort Study 1- Arm 2 vs Structured Interviews vs Cohort Study 2; Knowledge of sun protection score at baseline compared with score after completion of the arm. The hypothesis is that the focus group, usability test and structured interviews arms will not have significant change in knowledge. It is expected that cohort studies 1 and 2 will have significant change in knowledge of sun protection; Test type: Superiority; p < 0.1, Chi-squared

ADVERSE EVENTS:
Time Frame: 1 year
Description: Focus groups and structured interviews which involve talking with subjects have no risk of adverse medical events.
Groups:
- Cohort Study 1-arm 1: 31 subjects
  First cohort study: It is expected that each melanoma survivors will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants will be randomized to receive a survey item inviting selection of strategies to achieve sun-protected outdoor activities (structured goal attainment).
  Goal attainment: After reviewing daily UV exposure in the prior 10 days, participants will be randomized to structured (select strategies from a list of 7 items) or unstructured (submit a free text description of a strategy) goal attainment.
- Cohort Study 1-arm 2: 29 subjects each of 29 melanoma survivors in arm 2 will wear the sensor and transmit data for 21 days in the warm weather months of June-Aug 2019. It will take about 2 months to enroll the subjects. Subjects in both arms will receive daily text messages in a sequence starting with behavioral facilitation, outcome expectancies, self-efficacy, and self-regulation. On day 10, participants will receive a text message prompting review and reflection on the prior 10 days of UV exposure. Participants in arm 2 will be randomized to submit a free text description of their strategy (unstructured goal attainment).
Arm/Group | Focus Group | Usability Testing | Cohort Study 1-arm 1 | Cohort Study 1-arm 2 | Structured Interviews | Cohort Study 2
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/10 | 0/31 | 0/29 | 0/20 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/10 | 0/31 | 0/29 | 0/20 | 0/42
Other Adverse Events (participants affected / at risk) | 0/32 | 0/10 | 0/31 | 0/29 | 0/20 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT03344796/Prot_SAP_002.pdf
  • Informed Consent Form (2019-03-11): https://cdn.clinicaltrials.gov/large-docs/96/NCT03344796/ICF_001.pdf